CLINICAL TRIAL: NCT02875483
Title: Expedited Interval Tubal Scheduling: An Intervention to Increase Rates of Completion of Tubal Sterilization Within 6 Months Post-partum
Brief Title: Expedited Interval Tubal Scheduling
Acronym: ExITS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16D.494
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Female Tubal Sterilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Scheduling (Placebo Comparator): Group allocated to follow standard surgical scheduling practices
  Interventions: Other: Standard Scheduling
- Expedited Scheduling (Experimental): Group allocated to expedited scheduling practices
  Interventions: Other: Expedited Scheduling

INTERVENTIONS:
Other: Expedited Scheduling — Patients are scheduled for tubal ligation surgery prior to discharge from the post-partum hospital service, with target date 4-8 weeks post-partum.
  Arms: Expedited Scheduling
Other: Standard Scheduling — Scheduling of tubal surgery occurs after completion of post-partum office visit
  Arms: Standard Scheduling

SUMMARY:
Over 50% of all pregnancies that occur in the US are unintended, and unintended pregnancy is detrimental to maternal and child health. Tubal sterilization may be performed immediately following a delivery, or as an interval procedure remote from pregnancy. Many women request sterilization to follow delivery, but it is frequently not completed during the peri-partum hospitalization. Women who are denied an immediate post-partum tubal are generally candidates to complete the procedure as an interval surgery within a few months of delivery, but few do so. Women who request tubal sterilization and do not receive it are at highest risk for a rapid repeat pregnancy, with as many as 46% having an unintended pregnancy within 1 year.

The standard care at many institutions for a patient denied tubal sterilization during hospitalization is to offer a short term contraceptive and instruct the patient to follow up for the standard post-partum outpatient visit in 4-6 weeks. If the patient still desires tubal sterilization at that time, the surgical procedure will be scheduled. No-show rates for post-partum care are high at about 50%-60%, and therefore, many patients are never scheduled for their surgery. If the process of scheduling interval tubal sterilization surgery could be expedited, rates of completion could be improved.

DETAILED DESCRIPTION:
Identification of potential participants: On admission to the hospital for labor, all women will be asked if they were planning to tie their tubes after their delivery. Women who requested tubal ligation and have not received this on post-partum day one, and who are not anticipated to have it completed on post-partum days 2 or 3, and who did not have a contraceptive device (IUD or Nexplanon) placed that the time of delivery will be identified from hospital service lists.

Enrollment: All patients meeting inclusion criteria will be approached by study personnel and asked about whether sterilization is their preferred contraceptive method. If the potential participant still expresses a desire for permanent sterilization, the potential participant will be offered enrollment in the study. The study will be described, and the expected preferred method of sterilization identified. The participant will sign informed consent.

Allocation Concealment: A randomization sequence will be developed with a computerized number generator, and will generate participant assignments in a 1:1 ration with randomly permuted block sizes of 4, 6, and 8. A person not involved with study enrollment will place cards with participant assignments in a series of sequentially numbered, sealed opaque sealed envelopes. These envelopes will be stored on the post partum floor, and after a patient completes the informed consent, the next sequential envelope will be opened.

Randomization: The potential candidate will be randomized by opening of the next sequentially numbered sealed envelope. The assignment will be noted and disclosed. The assignment will be noted in the study chart, and the card with the assignment will be stored with the chart.

Study protocol following randomization:

If the participant is assigned to the standard care arm, the participant will be instructed to present for her post-partum visit, and that surgical procedure will be scheduled at that time. These participants will be offered appropriate short term contraceptive. This reflects current standard of care regarding post-partum follow up and contraception.

If the participant is assigned to the expedited scheduling arm, the preferred method of sterilization (laparoscopic or hysteroscopic) will be confirmed. The available dates for surgery in the appropriate window (4-8 weeks post-partum) will be offered, and the participant will confirm her preferred dates. The surgery scheduling team will be contacted, and the patient will be placed on the schedule. If a date cannot be definitively confirmed prior to discharge, the participant will be instructed to expect a call from the surgery schedulers to confirm the surgical date within 3 days of hospital discharge. In that phone call, administrators will provide information for pre-admission testing date to complete preoperative laboratory work if needed. The participant will be instructed to schedule a routine post-partum visit as well per usual protocols. All participants will be offered the appropriate short-term contraceptive.

Follow-up after hospital discharge. Patients in the expedited group will receive the standard phone calls from the surgery scheduling team regarding pre-operative appointments and the peri-operative nurses on the day prior to schedule surgery. Participants will not receive any other specialized reminders regarding their surgical date or intentions for follow up. If participants contact the office requesting a change to a surgical date, this will be allowed.

Per usual surgical procedures, if participants do not present for their scheduled surgery, they will be contacted and offered an opportunity to re-schedule. If participants miss more than one scheduled surgery date, they will not be contacted further to re-schedule; however, if the participant calls the office to schedule independently, another surgical date will be offered.

Patients in the standard of care group will receive standard discharge summary and instructions which include instruction to contact the outpatient OB-Gyn office to schedule post-partum follow-up in about 6 weeks. Once scheduled for an appointment, participants will receive the standard automated appointment reminder call or text. Participants will not receive any specialized reminders regarding follow-up for either routine post-partum care or regarding scheduling of sterilization surgery. Participants will not be seen by study personnel at this visit to encourage or facilitate scheduling of tubal, as the goal is for this group to receive current standard care. Data regarding the outcome of this visit will be abstracted from the post-partum chart by study personnel.

Study Completion:

Participants will be considered exited from the study at these endpoints:

* Tubal is completed as scheduled - do satisfaction survey: study complete
* Seen for follow up, and state definitively that they have changed mind about tubal and no longer desire it - do satisfaction survey: study complete (Survey B for survey specific to those who have changed their mind regarding tubal)
* Are seen for follow up within 6 month, state intention to complete tubal. It is done within 6 months. Do survey at time of tubal: study complete.
* Are seen for follow up within 6 months, state intention to complete tubal, but it has not been completed at 6 month mark - will be contacted by phone, queried about barriers and why not done, and complete satisfaction survey: study complete (Survey C for survey specific to non-completion of follow up)
* Are not seen for follow up at all within 6 months - will be contacted by phone at 6-month point to determine if tubal done elsewhere, method of contraception, interval pregnancy, complete satisfaction survey (Survey C): study complete

ELIGIBILITY:
Inclusion Criteria:

* >21 years of age (required for sterilization by Medicaid rules)
* Requested sterilization either during antepartum care or at time of delivery
* Did not have sterilization performed on L&D for any reason
* Confirmed desire for sterilization during post-partum hospitalization (has not changed mind)
* Has commercial or Medicaid insurance that will allow for outpatient surgery (including pregnancy-related emergency Medicaid)
* Consent to phone follow-up calls regarding study in the 6 months following enrollment

Exclusion Criteria:

* <21 years of age
* Unable to provide informed consent
* Not a candidate for a laparoscopic or hysteroscopic procedure for any medical reason
* Uninsured or undocumented status that would prevent scheduling of an outpatient surgery
* Unable to provide reasonably reliable contact information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
Completion of Tubal Sterilization | 6 months
  Proportion of participants who complete requested tubal ligation surgery within 6 months of their delivery.

SECONDARY OUTCOMES:
Participant Satisfaction | 6 months
  Participant satisfaction with process of scheduling and completing surgery
Repeat pregnancy Rates | 6 months
  Proportion of participants with rapid repeat pregnancy within 6 months of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mercier RJ, Perriera L, Godcharles C, Shaber A. Expedited Scheduling of Interval Tubal Ligation: A Randomized Controlled Trial. Obstet Gynecol. 2019 Dec;134(6):1178-1185. doi: 10.1097/AOG.0000000000003550. PMID 31764727